CLINICAL TRIAL: NCT06993285
Title: ADvanced ALzheimer Disease and Effects of Protologic and LAnguage Rehabilitation Tools (a Non-pharmacological Intervention) in Nursing Home.
Brief Title: ADvanced ALzheimer Disease and Effects of Protologic and LAnguage Rehabilitation Tools in Nursing Home (ADALPA)
Acronym: ADALPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laure JOLY, Professor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Central Hospital, Nancy France; Fondation Médéric Alzheimer (Other: Fondation Médéric Alzheimer)
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
Keywords: severe Alzheimer disease; non pharmacological intervention; protologic rehabilitation; speech therapist
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- return to communication verbally or non-verbally of patients with severe Alzheimer disease (Other): 9 patients over 60 years old with major neurocognitive disorders at an advanced stage, presenting behavioral disorders, no longer communicating, interacting and having little or no relationship with objects, with stereotyped behavior or apathy living in 3 nursing home will be recruted during 36 months.
  Each patient will receive a maximum of 34 weeks of Protologic and LAnguage adaptation rehabilitation by a speech therapist at a rate of one or two speech therapy sessions per week, for a total of 30 sessions maximum. All sessions are filmed and at posteriori analysed with the help of ELAN© software.
  Interventions: Other: Protologic and LAnguage adaptation rehabilitation

INTERVENTIONS:
Other: Protologic and LAnguage adaptation rehabilitation — Each patient will receive a maximum of 34 weeks of Protologic and LAnguage adaptation rehabilitation by a speech therapist at a rate of one or two speech therapy sessions per week, for a total of 30 sessions maximum. All sessions are filmed and at posteriori analysed with the help of ELAN© software

SUMMARY:
Background:

During Alzheimer's disease when cognitive disorders become too severe, language and communication are no longer present and/or mobilizable, and as a consequence there is a frequent discontinuation of Care and morever speech therapy rehabilitation. On this very specific subject of return to communication of patients suffering from very advanced Alzheimer's disease with cessation of communication, no data is currently avalable in the scientific literature to identify and define a "threshold for return to communication".

Objectives :

This study aims at obtaining a return to communication verbally (V) or non-verbally (NV), of patients living in nursing home suffering from severe neurocognitive disorders during Alzheimer disease using evaluation grids of V and NV communication.

Secondary objectives are the evaluation of recovery of a relationship with objects, quality of relashionship between patients and caregivers and family members , reduction in behavioral signs ( NPI-ES, EPADE survey), improved nutrition.

Method :

9 patients over 60 years old with major neurocognitive disorders at an advanced stage, presenting behavioral disorders, no longer communicating, interacting and having little or no relationship with objects, with stereotyped behavior or apathy living in 3 nursing home will be recruted during 36 months.

Each patient will receive a maximum of 34 weeks of Protologic and LAnguage adaptation rehabilitation by a speech therapist at a rate of one or two speech therapy sessions per week, for a total of 30 sessions maximum. All sessions are filmed and at posteriori analysed with the help of ELAN© software.

Attended results : The benefits of this research will be to objectivize an improvement in the cognitive state of patients, with a possible return to communication. Moreover, this study will provide a better understanding of neurocognitive disorders and their evolution after a Non-Pharmacological Intervention. The existence of improvements will also enable a change in the way caregivers and relatives look at these patients at an advanced stage, especially as at present, follow-up is generally discontinued as soon as language and communication are no longer present and can not be mobilized.

ELIGIBILITY:
Inclusion Criteria:

* subject aged ≥60 years
* living in nursing home
* presenting a neurocognitive disorder at an advanced stage
* MMSE <10
* NPI ES : presence of apathy and/or indifference and/or aberrant motor behavior
* subject having received oral information and representative having received complete information on the organization of the research and not having objected to the participation of the patient and to the exploitation of data
* Subject or representative having consented to the fixation, reproduction and exploitation of the audiovisual recording.

Exclusion Criteria:

* Delirium
* psychiatric disorder (diagnosed severe depressive disorder, diagnosed schizophrenia)
* Personnes benefiting from another non-pharmacological intervention or included in another research protocol
* subject deprived of liberty by a judicial or administrative decision

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Return to communication (YES / NO) during non pharmacological intervention | From enrollment to the end of non pharmacological intervention at 34 weeks
  The main objective is to authenticate a return to communication (YES / NO) during non pharmacological intervention sessions (maximum 30 sessions per patient) in patients for whom no communication existed at time 0 (each patient is his or her own witness). Authenticate according to the elements obtained from the communication observation grids non-verbal (NV) and verbal (V).

CONTACTS AND LOCATIONS:
Overall Officials: Laure JOLY, Professor, Study Director — Central Hospital, Nancy, France; Clotilde Caillet-Gipeaux, Principal Investigator
Locations (1):
- CentralHNF, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
Under the responsibility of the promoter or in application of specific legal or regulatory provisions, the categories of persons described below have access to data processed, within the limits of their authorizations with regard to their functions and under conditions that comply with regulations.
  These categories of persons are bound by professional secrecy under the conditions defined by articles 226-13 and 226-14 of the French penal code.
  Recipients of indirectly identifying data concerning individuals participating in the research
  * the sponsor and individuals or legal entities acting on its behalf;
  * principal investigators;
  * professionals involved in the research and staff acting under their responsibility or authority (investigator, IRC, CRA, TEC of the investigating center )
  * staff of companies in the group to which the sponsor belongs and whose participation is necessary for data processing within the framework of the research;
  * healthcare professionals involved
Supporting Information: Study Protocol, CSR
Time Frame: 2030
Access Criteria: Data may be transmitted to companies in the group to which the promoter belongs and to its contractual part All data and information concerning the person taking part in the research will remain strictly confidential. Persons with direct access to these data and information in accordance with the legislative and regulatory provisions in force, in particular articles L.1121-3 and R.5121-13 of the French Public Health Code take all necessary precautions to ensure the confidentiality of information relating to the experimental products, the research, the persons taking part in it and the results obtained.
  In accordance with article R.5121-13 of the French Public Health Code, these persons may, without the sponsor's consent, provide information relating to research only to the Minister for Health, medical public health inspectors, pharmacist public health inspectors, the Director General and inspectors of the French National Agency for the Safety of Medicines and Health Products.

REFERENCES:
- See also: The aims of this project are to improve verbal and non-verbal communication among residents of nursing homes living with advanced Alzheimer's disease and to enable them interaction and communication. — https://lnkd.in/eeZ2jbgU